CLINICAL TRIAL: NCT06313567
Title: Metronomic Capecitabine as Adjuvant Therapy in Stage III Gastric Cancer: a Multicentre, Open-label, Parallel-group, Randomised, Controlled, Phase 3 Trial
Brief Title: Metronomic Capecitabine in Stage III Gastric Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Dazhi Xu, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Meca-GC
Record Dates: First submitted 2024-03-10; First posted 2024-03-15 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Gastric Cancer
Keywords: Gastric Cancer; Metronomic capecitabine
MeSH Terms: conditions — Stomach Neoplasms | interventions — Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metronomic capecitabine (Experimental): Low-dose capecitabine maintenance (500 mg/m2 body surface area twice daily for 1 year) after completion of standard adjuvant chemotherapy,
  Interventions: Drug: Metronomic capecitabine group
- Standard therapy group (Active Comparator): Observation after completion of standard adjuvant chemotherapy,
  Interventions: Other: Observation

INTERVENTIONS:
Drug: Metronomic capecitabine group — 500 mg/m2 body surface area twice daily for 1 year; metronomic capecitabine group
  Arms: Metronomic capecitabine
Other: Observation — observation
  Arms: Standard therapy group

SUMMARY:
The purpose of this study is to find out whether treatment with metronomic capecitabine will improve the survival of gastric cancer patients with stage III who had received standard treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Lower age limit of research subjects 18 years old and upper age limit of 80 years old.
2. Be proven to be primary adenocarcinoma of gastric cancer and staged III by pathological evidences
3. R0 gastrectomy with D2 lymphadenectomy
4. ECOG (ECOG score standard) performance status of 0 or 1 and expected to survive more than 6 months
5. No contraindications, including normal peripheral blood routine, liver and kidney function and electrocardiogram （WBC≥3.5 x 109 /L, NEU≥1.2 x 109 /L,PLT≥90 x 109 /L and HGB≥80g/L).

Exclusion Criteria:

1. History of chemotherapy, radiotherapy, immunotherapy or target therapy
2. Multiple primary tumors
3. Suffering from other serious diseases, including cardiovascular, respiratory, kidney, or liver disease, complicated by poorly controlled hypertension, diabetes, mental disorders or diseases
4. Unavailable for R0 resection and D2 lymph node dissection.
5. Patients with stage IV gastric cancer

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 722 (Estimated)
Dates: Start 2024-03-10 (Actual); Primary Completion 2029-03-10 (Estimated); Study Completion 2029-03-10 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 3-year
  DFS

SECONDARY OUTCOMES:
Overall survival | 3-year
  OS
Side effects | 1-year
  Complications such as Nausea, vomiting, myelosuppression and Liver or kidney function disorder

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided